CLINICAL TRIAL: NCT01025934
Title: Intravitreal Bevacizumab for Surgical Treatment of Severe Proliferative Diabetic Retinopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: Napoli CTO Hospital (Unknown)
Purpose: Treatment
Other Study IDs: IVBDRNA
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2009-12-04 (Estimated); Status verified 2009-12

CONDITIONS: Proliferative Diabetic Retinopathy
MeSH Terms: interventions — Bevacizumab; salicylhydroxamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 7 days (Active Comparator)
  Interventions: Drug: Bevacizumab
- 20 days (Active Comparator)
  Interventions: Drug: Bevacizumab
- sham (Sham Comparator)
  Interventions: Other: sham

INTERVENTIONS:
Drug: Bevacizumab
  Arms: 20 days; 7 days
Other: sham
  Arms: sham

SUMMARY:
The purpose of this study is to evaluate the role, the safety and the effectiveness of Intravitreal Bevacizumab injections as an adjunct to vitrectomy in the management of severe proliferative diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* vitreous haemorrhage
* tractional retinal detachment
* active proliferative diabetic retinopathy.

Exclusion Criteria:

* neovascular glaucoma
* cataract
* combined traction and rhegmatogenous RD

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult

REFERENCES:
- [Derived] di Lauro R, De Ruggiero P, di Lauro R, di Lauro MT, Romano MR. Intravitreal bevacizumab for surgical treatment of severe proliferative diabetic retinopathy. Graefes Arch Clin Exp Ophthalmol. 2010 Jun;248(6):785-91. doi: 10.1007/s00417-010-1303-3. Epub 2010 Feb 5. PMID 20135139